CLINICAL TRIAL: NCT00689845
Title: A Clinico-Pathologic Study of Primary Mediastinal B-Cell Lymphoma (IELSG 26)
Brief Title: Combination Chemotherapy and Rituximab in Treating Patients With Primary Mediastinal Diffuse Large B-Cell Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000588011; USCTU-IELSG-26-RHM-CAN0546; EU-20818; EudraCT 2006-005794-22; USCTU-07/Q1704/68
Record Dates: First submitted 2008-06-03; First posted 2008-06-04 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Bleomycin; Filgrastim; Rituximab; Cyclophosphamide; Cytarabine; Doxorubicin; etoposide phosphate; Ifosfamide; Methotrexate; Prednisolone; Prednisone; Vincristine; Vindesine

ARMS (5):
- Cohort 1 (Experimental): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1. Patients also receive oral prednisolone on days 1-5. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisolone; Drug: vincristine sulfate
- Cohort 2 (Experimental): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1, oral prednisolone on days 1-5, and filgrastim (G-CSF) subcutaneously (SC) on days 5-12. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisolone; Drug: vincristine sulfate
- Cohort 3 (Experimental): Patients receive rituximab IV on days 1, 22, 43, 64, 85, and 106; cyclophosphamide IV and doxorubicin hydrochloride IV on days 1, 15, 29, 43, 57, and 71; methotrexate IV on days 8, 36, and 64; vincristine IV on days 8, 22, 36, 50 ,64, and 78; bleomycin IV on days 22, 50, and 78; and oral prednisolone on days 1-84, followed by a taper.
  Interventions: Biological: bleomycin sulfate; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: methotrexate; Drug: prednisolone; Drug: vincristine sulfate
- Cohort 4 (Experimental): Patients receive rituximab IV on days 1, 22, 43, 64, 85, and 106; cyclophosphamide IV on days 1, 29, and 57; doxorubicin hydrochloride IV on days 1, 15, 29, 43, 57, and 71; etoposide phosphate IV on days 15, 16, 43, 44, 71, and 72; vincristine IV and bleomycin IV on days 8, 22, 36, 50, 64, and 78; and oral prednisolone on days 1-84, followed by a taper.
  Interventions: Biological: bleomycin sulfate; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide phosphate; Drug: prednisolone; Drug: vincristine sulfate
- Cohort 5 (Experimental): Patients receive rituximab IV, doxorubicin hydrochloride IV, and cyclophosphamide IV on day 1; vindesine IV and bleomycin IV on days 1 and 5; oral prednisone on days 1-5; methotrexate intrathecally on day 2; and G-CSF SC on days 6-13 for 4 courses in the absence of disease progression or unacceptable toxicity. After completion of 4 courses of R-ACVBP, patients receive consolidation therapy comprising high-dose methotrexate IV, rituximab IV, ifosfamide IV, etoposide phosphate IV, and cytarabine SC according to protocol GELA LNH03-2B.
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: cytarabine; Drug: doxorubicin hydrochloride; Drug: etoposide phosphate; Drug: ifosfamide; Drug: methotrexate; Drug: prednisone; Drug: vindesine

INTERVENTIONS:
Biological: bleomycin sulfate — Given IV
  Arms: Cohort 3; Cohort 4; Cohort 5
Biological: filgrastim — Given subcutaneously
  Arms: Cohort 2; Cohort 5
Biological: rituximab — given IV
Drug: cyclophosphamide — Given IV
Drug: cytarabine — Given subcutaneously
  Arms: Cohort 5
Drug: doxorubicin hydrochloride — Given IV
Drug: etoposide phosphate — Given IV
  Arms: Cohort 4; Cohort 5
Drug: ifosfamide — Given IV
  Arms: Cohort 5
Drug: methotrexate — Given IV
  Arms: Cohort 3; Cohort 5
Drug: prednisolone — Given orally
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: prednisone — Given orally
  Arms: Cohort 5
Drug: vincristine sulfate — Given IV
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: vindesine — Given IV
  Arms: Cohort 5

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving rituximab together with one of five different combination chemotherapy regimens may kill more cancer cells.

PURPOSE: This clinical trial is studying giving rituximab together with combination chemotherapy to see how well it works in treating patients with primary mediastinal diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To systematically analyze the phenotype and molecular characteristics in patients with primary mediastinal diffuse large B-cell lymphoma.
* To determine the PET response rate following chemoimmunotherapy in these patients.

Secondary

* To obtain data, on a nonrandomized basis, regarding the outcomes of treatment using different chemoimmunotherapy regimens and using or omitting mediastinal radiotherapy, depending upon the practice of the participating institutions.
* To analyze progression-free and overall survival in patients treated with these regimens.

OUTLINE: This is a multicenter study.

Patients receive any one of the following standard chemoimmunotherapy regimens.

* Cohort 1 (R-CHOP-21): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1 and oral prednisolone on days 1-5. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Cohort 2 (R-CHOP-14): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1, oral prednisolone on days 1-5, and filgrastim (G-CSF) subcutaneously (SC) on days 5-12. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
* Cohort 3 (R-MACOP-B): Patients receive rituximab IV on days 1, 22, 43, 64, 85, and 106; cyclophosphamide IV and doxorubicin hydrochloride IV on days 1, 15, 29, 43, 57, and 71; methotrexate IV on days 8, 36, and 64; vincristine IV on days 8, 22, 36, 50 ,64, and 78; bleomycin IV on days 22, 50, and 78; and oral prednisolone on days 1-84, followed by a taper.
* Cohort 4 (R-VACOP-B): Patients receive rituximab IV on days 1, 22, 43, 64, 85, and 106; cyclophosphamide IV on days 1, 29, and 57; doxorubicin hydrochloride IV on days 1, 15, 29, 43, 57, and 71; etoposide phosphate IV on days 15, 16, 43, 44, 71, and 72; vincristine IV and bleomycin IV on days 8, 22, 36, 50, 64, and 78; and oral prednisolone on days 1-84, followed by a taper.
* Cohort 5 (R-ACVBP): Patients receive rituximab IV, doxorubicin hydrochloride IV, and cyclophosphamide IV on day 1; vindesine IV and bleomycin IV on days 1 and 5; oral prednisone on days 1-5; methotrexate intrathecally on day 2; and G-CSF SC on days 6-13 for 4 courses in the absence of disease progression or unacceptable toxicity. After completion of 4 courses of R-ACVBP, patients receive consolidation therapy comprising high-dose methotrexate IV, rituximab IV, ifosfamide IV, etoposide phosphate IV, and cytarabine SC according to protocol GELA LNH03-2B.

Patients with an International Prognostic Index score of 4 or greater or disease in close proximity to the spinal cord or cerebral meninges may receive prophylactic treatment to the CNS according to local protocol.

Beginning 8 weeks after completion of chemoimmunotherapy, patients undergo radiotherapy to the original tumor volume according to local protocol.

Fresh or fixed tissue from prior biopsy is obtained if possible. Samples are analyzed for CD3, CD20, CD30, CD15, CD10, Bcl-6, Bcl-2, MAL protein (if available), and Ki-67 via immunohistochemistry.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary mediastinal diffuse large B-cell lymphoma

  * CD20-positive disease
  * Any stage of disease
  * Must have a dominant mass within the anterior mediastinum

PATIENT CHARACTERISTICS:

* ANC ≥ 1.5 x 10^9/L (unless due to lymphoma)
* Platelets ≥ 100 x 10^9/L (unless due to lymphoma)
* WBC ≥ 3.0 x 10^9/L (unless due to lymphoma)
* Serum creatinine ≤ 2 times upper limit of normal (ULN) (unless due to lymphoma)
* AST/ALT ≤ 2.5 times ULN (unless due to lymphoma)
* Total bilirubin ≤ 2.5 times ULN (unless due to lymphoma)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be fit to receive chemotherapy with curative intent
* No evidence of clinically significant cardiac disease* within the past 12 months, including any of the following:

  * Symptomatic ventricular arrhythmias
  * Congestive heart failure
  * Myocardial infarction NOTE: * Cardiac compromise due to local extension of lymphoma will not be an exclusion criterion in the absence of other cardiac disease.
* No known HIV infection
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Able and willing to give informed consent and to undergo staging, including PET scanning

PRIOR CONCURRENT THERAPY:

* No prior treatment for lymphoma
* Prior corticosteroids for up to 1 week allowed for the relief of local compressive symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-06

PRIMARY OUTCOMES:
Complete response rate on PET scanning at the completion of chemoimmunotherapy

SECONDARY OUTCOMES:
Progression-free survival
Death
Survival time

CONTACTS AND LOCATIONS:
Overall Officials: Peter Johnson, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (8):
- United Kingdom (8):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - St. George's Hospital, London, England
  - Christie Hospital, Manchester, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Saint Bartholomew's Hospital, London